CLINICAL TRIAL: NCT07125209
Title: Cognitive Impact of Neoadjuvant Chemotherapy for Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-1115; SMPH/OB-GYN/GYN ONCOLOGY (Other: UW Madison); Protocol Version 7/23/25 (Other: UW Madison); UW25061 (Other: OnCore ID)
Record Dates: First submitted 2025-08-07; First posted 2025-08-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer; Cognitive Change
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — optional blood draw for research purposes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Receiving Neoadjuvant Chemotherapy for Ovarian Cancer
  Interventions: Other: Patient Reported Outcomes Assessment; Other: Cognitive and General Health Assessments

INTERVENTIONS:
Other: Patient Reported Outcomes Assessment — Functional Assessment of Cancer Therapy - Ovarian (FACT-O) and Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) will be used to assess patient reported outcomes.
  Other Names: FACT-O; FACT-Cog
Other: Cognitive and General Health Assessments — * Rey Verbal Learning Test
  * Trail Making Test
  * Patient Health Questionnaire (PHQ-2)
  * Mini Mental State Exam (MMSE)
  * Controlled Oral Word Association Test of the Multilingual Aphasia Examination

SUMMARY:
The purpose of this research is to assess several components of cognition in patients recently diagnosed with advanced epithelial ovarian cancer and who will be undergoing neoadjuvant chemotherapy for treatment of the cancer. 18 participants will be enrolled and can expect to be on study for approximately 10 months.

DETAILED DESCRIPTION:
Participants undergoing neoadjuvant chemotherapy for newly diagnosed, advanced epithelial ovarian cancer will be assessed for patient reported outcomes (including subjective cognitive impairment) and objective cognitive function at baseline, following three cycles of neoadjuvant chemotherapy, at the completion of adjuvant chemotherapy or transition to alternate treatment regimen for patients who progress through primary treatment, and six months following treatment completion. Patient reported outcomes will be assessed using the FACT-O and subjective cognitive impairment will be assessed using the FACT-Cog surveys.

The NCCN distress thermometer is used to screen for distress levels routinely in the gynecologic oncology clinic. For those who complete this screening as part of their clinical care, those results will also be used as a quality of life measure. The cognitive domains of learning and memory, processing speed, and executive function will be assessed using the Rey Verbal Learning Test, Trail Making Test, and the Controlled Oral Word Association of the Multilingual Aphasia Examination, as recommended by the International Cognition and Cancer Task force for studies of cognition in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Pathological diagnosis of suspected epithelial ovarian cancer; of note, patients with suspected epithelial ovarian cancer who are pending a pathological diagnosis/biopsy may be enrolled onto the study ahead of their biopsy. If the biopsy result is later inconsistent with epithelial ovarian cancer, they will be removed from the study and replaced
* Planned to received neoadjuvant chemotherapy with carboplatin and paclitaxel; alternatives to these agents including abraxane, docetaxel, cisplatin may be used if patients have a chemotherapy reaction or otherwise cannot receive carboplatin and paclitaxel per usual standard of care
* Patients may be receiving bevacizumab and may receive PARP inhibitors as a maintenance treatment; those receiving any other targeted therapy will be excluded

Exclusion Criteria:

* History of diagnosed cognitive impairment, including dementia
* History of traumatic brain injury
* English is not their primary language
* Known hearing or visual impairment not corrected with hearing devices and glasses/contacts
* Upper extremity motor impairment that would impact ability to perform the Trail Making Test
* Baseline Mini Mental State Exam (MMSE) score less than 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants scheduled to receive neoadjuvant chemotherapy for treatment of ovarian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The Mini Mental State Exam (MMSE) | baseline, after 3 cycles of neoadjuvant chemotherapy (up to 2 months), after completion of adjuvant therapy (up to 4 months), and 6 months following treatment (up to 10 months on study)
  The MMSE is a common overall test of cognition used in research and clinical settings. It is an 11 item test that assesses five domains of cognition: orientation, registration, attention, recall and language. This measure takes around 5-10 minutes to complete and is scored out of 30 with scores of 18-23 representing mild cognitive impairment and scores of 17 or less representing severe cognitive impairment.

SECONDARY OUTCOMES:
Controlled Oral Word Association Test (COWAT) | baseline, after 3 cycles of neoadjuvant chemotherapy (up to 2 months), after completion of adjuvant therapy (up to 4 months), and 6 months following treatment (up to 10 months on study)
  Participant is asked to list as many words (other than people's names or places) beginning with a specific letter as they can in one minute. Number of unique words that qualify are counted.
Trail Making Test (TMT) Parts A and B | baseline, after 3 cycles of neoadjuvant chemotherapy (up to 2 months), after completion of adjuvant therapy (up to 4 months), and 6 months following treatment (up to 10 months on study)
  The TMT is a test of complex attention. Part A asks participants to connect circles on a page containing the numbers 1-25 in ascending order. Part B asks participants to connect circles containing the numbers 1-13 and the letters A-L in alternating ascending order (eg: 1, A, 2, B, etc). These tests are timed and a participant's score is the amount of time it takes to complete the entire task for each part; errors do not incur a score penalty but contribute to the overall time to complete the task. This takes approximately 5-10 minutes to complete
Patient Health Questionnaire-2 (PHQ-2) | baseline, after 3 cycles of neoadjuvant chemotherapy (up to 2 months), after completion of adjuvant therapy (up to 4 months), and 6 months following treatment (up to 10 months on study)
  The PHQ2 is a two item screening test that asks about the frequency of depressed mood and anhedonia over the past two weeks. Subjects whose answers receive a score of three or greater (on a scale of 0-6) are considered to be at risk for depression and should undergo further evaluation. This screening test takes around one minute to administer.
Functional Assessment of Cancer Therapy - Ovarian (FACT-O) | baseline, after 3 cycles of neoadjuvant chemotherapy (up to 2 months), after completion of adjuvant therapy (up to 4 months), and 6 months following treatment (up to 10 months on study)
  The FACT-O is a validated and commonly used quality of life assessment utilized in many clinical research studies that assess 39 items/symptoms common amongst cancer patients generally with items included that are specifically common amongst ovarian cancer patients, including questions related to gastrointestinal symptoms and sexual health. Total scores range from 0 - 156 with higher scores indicative of better quality of life.
Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) | baseline, after 3 cycles of neoadjuvant chemotherapy (up to 2 months), after completion of adjuvant therapy (up to 4 months), and 6 months following treatment (up to 10 months on study)
  The FACT-Cog is a patient reported outcomes measure assessing 37 cognitively-related symptoms, as well as their perceived impact on quality of life from the past 7 days. Scoring is from 0-4 in each of the following domains: perceived cognitive impairments, comments from others, perceived cognitive abilities, impact on quality of life. Total scores range from 0 -148 with higher scores indicating better perceived cognitive functioning.
Rey Auditory Verbal Learning Test (RAVLT) | baseline, after 3 cycles of neoadjuvant chemotherapy (up to 2 months), after completion of adjuvant therapy (up to 4 months), and 6 months following treatment (up to 10 months on study)
  The RAVLT is a test of immediate memory and verbal learning where participants are given three trials to recall as many words as possible from a 15-item list. Participants are asked to repeat this list one additional time after a 5-25 minute delay. This takes around 4 minutes to complete. Number of correct words from the list of 15 are reported for each trial.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Barroilhet, MD, Principal Investigator — UW Carbone Cancer Center
Locations (1):
- UW Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No